CLINICAL TRIAL: NCT03627598
Title: High Flow Nasal Oxygen in Addition to Non Invasive Ventilation During Hypercapnic Respiratory Failure
Brief Title: High Flow Oxygen and Non Invasive Ventilation for Hypercapnic Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Nejla Tilouche, medecine doctor, University Hospital, Mahdia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140284
Record Dates: First submitted 2018-08-04; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Hypercapnic Respiratory Failure
Keywords: high flow oxygen; non invasive ventilation; hypercapnic respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Reference Standards

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard group (Active Comparator): NIV alternating with low oxygen therapy at 1 to 4 liters per minute to obtain SpO2 between 88% and 94%.
  Interventions: Device: standard
- HFNC group (Experimental): NIV alternating with HFNC delivering the equivalent inspired fraction of oxygen (FiO2) with a flow at 30 to 60 liters/min through an Optiflow nasal interface.
  Interventions: Device: HFNC

INTERVENTIONS:
Device: HFNC — patients will receive high flow warmed air with low inspired fraction of oxygen between non invasive ventilation sessions
  Arms: HFNC group
Device: standard — patients will receive low flow oxygen therapy at 1 to 4 liters per minute
  Arms: standard group

SUMMARY:
this study evaluates high flow oxygen therapy in addition to non invasive ventilation (NIV) to treat hypercapnic respiratory failure. Between sessions of NIV, half of participants will have high flow nasal cannula while the others will have standard low flow oxygen therapy.

DETAILED DESCRIPTION:
High Flow Nasal Cannula (HFNC) is a new way of oxygen therapy that has gained interest in the management of patients with acute respiratory failure. It allows reaching a high flow air up to 60 liters / min via a nasal cannula with a humidification and warming of the air administered. It has a number of physiological effects such as wash out of anatomical dead space, generation of a small PEEP and high inspired fraction of oxygen which enhances compliance and reduces inspiratory efforts.

NIV is the corner stone in the treatment of severe COPD exacerbation. Nevertheless, prolonged application of the facial mask expose to local complications and intolerance which can be a cause of failure, so reducing the duration of exposure to this procedure is important.

The role of HFNC in supplementing NIV effect during hypercapnic respiratory failure has not been assessed. Much of the data available on HFNC are about hypoxemic respiratory failure.

Because of its physiological effects, it can be hypothesized that HFNC in addition to NIV can shorten its duration by facilitating carbon dioxide clearance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years with a diagnosis of acute-on-chronic respiratory failure and respiratory acidosis requiring NIV.

Exclusion Criteria:

* Patient included in another study
* Patients intubated at ICU admission or within 12 hours
* Contraindication to NIV including: pneumothorax, Hemodynamic instability, GCS less than 12, facial malformation
* Asthma
* A do not intubate order
* Neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
duration of NIV | 28 days
  number of days patients received NIV, and for patients with home NIV: it is the number of days spent to achieve the usual daily NIV hours with clinical and gasometric stability

SECONDARY OUTCOMES:
Time to obtain NIV withdrawal criteria | 28 days
  the day patients do not have signs of acute respiratory failure and no respiratory acidosis (pH <7.36)
NIV failure | 28 days
  need for intubation or death
ICU length of stay | 28 days
  number of days spent in the ICU for this episode of exacerbation
ICU Mortality | 28 days
  death in the ICU during the recorded episode

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit, Mahdia, Tunisia

REFERENCES:
- [Background] Lepere V, Messika J, La Combe B, Ricard JD. High-flow nasal cannula oxygen supply as treatment in hypercapnic respiratory failure. Am J Emerg Med. 2016 Sep;34(9):1914.e1-2. doi: 10.1016/j.ajem.2016.02.020. Epub 2016 Feb 12. No abstract available. PMID 26947372
- [Result] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908